CLINICAL TRIAL: NCT07361861
Title: The Effects of Hyperbaric Oxygen Therapy at Intermediate Pressure (1.75 ATA) on VO₂ Max and Inflammatory Cytokine Profiles
Brief Title: Evaluating Whether Hyperbaric Oxygen Therapy Can Improve VO₂-Max and Reduce Inflammation Markers in Healthy Adults Ages 30-60.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, John Powers, Principal Investigator, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00007903
Record Dates: First submitted 2026-01-21; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Fitness; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hyperbaric Oxygen Therapy 1.75 atmospheres (Experimental): Will complete 24 HBOT sessions, each lasting 100 minutes, over 8 weeks.
  Interventions: Device: Hyperbaric Oxygen Therapy

INTERVENTIONS:
Device: Hyperbaric Oxygen Therapy — 24 Hyperbaric Oxygen Therapy, each lasting 100 minutes, 3 times a week for 8 weeks.

SUMMARY:
The purpose of this study is to determine whether hyperbaric oxygen therapy (HBOT) at 1.75 atmospheres of pressure (ATA) improves cardiovascular fitness (VO₂ max) and reduces inflammation in healthy adults. HBOT involves breathing pure oxygen in a pressurized chamber and is considered investigational for this use.

Recent research has shown that different HBOT pressures can have different effects on inflammation. Specifically, some inflammatory cytokines (measurable markers of inflammation in the body) appear to decrease at low pressures like 1.3 ATA, while a different set of cytokines responds better at higher pressures, such as 2.0 ATA.

Cytokines are small proteins that play a crucial role in cell signaling, particularly within the immune system. They help regulate inflammation, infection response, and overall immune function. While some cytokines promote inflammation to fight off threats, others help reduce inflammation when it's no longer needed. An imbalance in cytokines - especially excessive inflammatory cytokines - can contribute to chronic inflammation, cardiovascular disease, and other health issues.

In this study, we are testing an intermediate pressure - 1.75 ATA - to see if we can target both sets of cytokines at once. If successful, this approach could offer broader anti-inflammatory benefits.

We are also interested in how this intermediate pressure may improve VO₂ max, a key indicator of cardiovascular fitness. Since VO₂ max is strongly linked to heart health and overall longevity, finding a safe and effective way to improve it has meaningful implications not just for athletes, but for anyone looking to enhance their fitness and well-being.

ELIGIBILITY:
Inclusion Criteria:

* physically active individuals with no history of chronic illness or HBOT exposure within the last three months.

Exclusion Criteria:

* individuals with contraindications to HBOT, including lung diseases or claustrophobia.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Cytokine levels | From enrollment to 4 weeks after the end of treatment (12 weeks after first treatment).
  Cytokines will be measured via blood analysis. Samples will be taken before treatment, at the midpoint, at the end, and 4 weeks post treatment. This is a measure of inflammation in the body.
VO2 max testing | From enrollment to 4 weeks post treatment (12 weeks after first treatment)
  A treadmill VO2 max test measured before treatment, at treatment midpoint, at the end of treatment, and 4 weeks after conclusion of treatment. This is an indicator of cardiovascular health.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - ATX Hyperbarics, Austin, Texas
  - Westlake Medical Arts, Austin, Texas

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2025-12-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT07361861/Prot_000.pdf